CLINICAL TRIAL: NCT03163992
Title: Pembrolizumab in HCC
Brief Title: Pembrolizumab in Advanced Hepatocellular Carcinoma as Second-line Treatment After Failure of Sorafenib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12-127
Record Dates: First submitted 2017-04-26; First posted 2017-05-23 (Actual); Results first posted 2022-08-04 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Pembrolizumab (MK-3475) 200 mg every 3 weeks (Q3W)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- pembrolizumab (Experimental): Pembrolizumab (MK-3475) 200 mg every 3 weeks (Q3W)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (MK-3475) 200 mg every 3 weeks (Q3W)
  Other Names: MK3475

SUMMARY:
This is a single-arm, single-center, open-label trial of pembrolizumab (MK-3475) in subjects with advanced hepatocellular carcinoma as second-line treatment after failure of sorafenib.

Approximately 60 subjects will be enrollment to evaluate the efficacy and safety of pembrolizumab.

Enrollment will begin with all subjects without regard for PD-L1 expression status.

An evaluable specimen for PD-L1 status must be available and confirmed prior to enrollment.

All study subjects will be evaluated every 6 weeks (+/- 7 days) following the date of IP drug adminstration for the first 12 months and every 12 weeks (+/- 7 days) thereafter until progression of disease is documented with radiologic imaging (computed tomography or magnetic resonance imaging).

The primary efficacy endpoint is ORR (objective response rate) per RECIST 1.1.

DETAILED DESCRIPTION:
Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final contact. After a screening phase of up to 28 days, eligible subjects will receive treatment beginning on Day 1 of each 3week dosing cycle for pembrolizumab.

Treatment with pembrolizumab will continue until documented disease progression, unacceptable adverse event(s),intercurrent illness that prevents further administration of treatment, investigators' decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, subject receives 24 months of pembrolizumab, or administrative reasons requiring cessation of treatment. After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events and events of clinical interest will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier).

Subjects who discontinue after 24months of therapy for reasons other than disease progression or intolerability or who discontinue after attaining a CR may be eligible for up to one year of retreatment after they have experienced radiographic disease progression.

Subjects who discontinue for reasons other than disease progression will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone for overall survival until death, withdrawal of consent, or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent for Biomedical Research. However, the subject may participate in the main trial without participating in Biomedical Research.
2. Have histologically or cytologically confirmed diagnosis of HCC (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible) based on pathology report.
3. Have Barcelona Clinic Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach.
4. Have a Child-Pugh class A liver score
5. Has experienced documented objective radiographic or clinical disease progression during first-line sorafenib therapy.
6. Have measurable disease based on RECIST1.1 as determined by investigator.
7. Be willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality for assessment of biomarker status. Repeat samples may be required if adequate tissue is not provided. Newly obtained endoscopic biopsy specimens are preferred to archived samples and formalin-fixed, paraffin-embedded (FFPE) block specimens are preferred to slides.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has received sorafenib within 14 days of first dose of study medication.
3. Has had esophageal or gastric variceal bleeding within the last 6 months. All subjects will be screened for esophageal varices, unless such screening has been performed in the past 12 months before first dose of treatment. If varices are present, they should be treated according to institutional standards before starting study treatment.
4. Had a solid organ transplant.
5. Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
7. Has received locoregional therapy to liver (transcatheter chemoembolization [TACE], transcatheter embolization [TAE], radiation, radioembolization, or ablation) or major surgery to liver or other site within 4 weeks prior to the first dose of study drug. Minor surgery (e.g., simple excision, tooth extraction) must have occurred at least 7 days prior to the first dose of study treatment (Cycle 1, Day 1).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient enrollment date was 26 Dec 2017 and the last patient enrollment date was 11 Jun 2019.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 60
Completed | 1
Not Completed | 59

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 32
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 60
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity. (biomarker negative vs biomarker Advanced Hepatocellular Carcinoma)
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI Complete Response (CR); Disappearance of all target lesions Partial Response (PR); >=30% decrease in the sum of the longest diameter of target lesions Overall Response (OR) = CR + PR
Time Frame: through study completion, an average of 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
Participants
  PR | 6
  SD | 30
  PD | 17
  CR | 0
  NA | 7

2. Secondary Outcome: Progression-free Survival (PFS) and Overall Survival (OS)
Description: Progression-free survival (PFS) was defined as the time from the started of treatment until the date of disease progression or death resulting from any cause.
  Overall survival was measured from the started of treatment to the date of death from any cause.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  Progression-free survival (PFS) is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Time Frame: through study completion, an average of 24 months
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
months
  PFS | 2.8 [2.6 to 4.7]
  OS | 8.3 [5.4 to 10.9]

ADVERSE EVENTS:
Time Frame: 2 year
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 35/60
Serious Adverse Events (participants affected / at risk) | 8/60
Other Adverse Events (participants affected / at risk) | 24/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=60)
fatigue (General disorders) | 8 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=60)
pruritis (Skin and subcutaneous tissue disorders) | 5 (5)
diarrhea (Gastrointestinal disorders) | 4 (4)
constipation (Gastrointestinal disorders) | 2 (2)
elevated liver enzyme (Hepatobiliary disorders) | 6 (6)
hyperbilirubinemina (Hepatobiliary disorders) | 5 (5)
hyperthyroidism (Endocrine disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03163992/Prot_SAP_000.pdf